CLINICAL TRIAL: NCT06474819
Title: Left Septal or Deep Septal Pacing to Prevent Pacing-induced Cardiomyopathy
Acronym: DEEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut d'Investigació Biomèdica de Bellvitge (Other)
Collaborators: Fundació La Marató de TV3 (Other); Hospital Universitari de Bellvitge (Other)
Responsible Party: Principal Investigator, Andrea Di Marco, Principal Investigator, Institut d'Investigació Biomèdica de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DEEP
Record Dates: First submitted 2024-06-19; First posted 2024-06-26 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Complete Heart Block; Second Degree Atrioventricular Block Möbitz Type II

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- deep (Experimental): The ventricular lead will be penetrated into the basal interventricular septum aiming at left septal pacing and, if not possible, at least deep septal pacing with a paced QRS duration <=140ms.
  Interventions: Device: Pacemaker implant
- Apex (Active Comparator): The ventricular lead will be placed in the right ventricular apex.
  Interventions: Device: Pacemaker implant

INTERVENTIONS:
Device: Pacemaker implant — All patients in the study will have a clear indication for a permanent pacemaker. The type of device (single or dual chamber) will be chosen as per clinical practice. The only difference between the two groups of the study will be the position of the ventricular lead.

SUMMARY:
Multicenter randomized controlled trial which will include patients with left ventricular ejection fraction >50% requiring a first implant of a cardiac pacemaker with expected high pacing percentages.

Patients will be randomized 1:1 to right ventricular apical pacing vs left septal or deep septal pacing. The primary endpoint will be pacing-induced cardiomyopathy during the first year of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* First implant of a single-chamber or dual chamber pacemaker due to persistent bradycardia associated with high degree atrio-ventricular (AV) block (complete AV block or second degree type II AV block), with second-degree type I AV block (symptomatic or associated with intra-hisian or infra-hisian block), or with atrial fibrillation with symptomatic slow ventricular rate (<45lpm).
* LVEF>50% at echocardiography performed maximum 7 days before pacemaker implant.
* Informed consent signature.

Exclusion Criteria:

* Life expectancy <12 months
* Severe cardiac valvular abnormality requiring intervention
* Unstable Angina, Acute myocardial infarction, coronary revascularization, valvular surgery or valvular percutaneous intervention in the 90 days prior to pacemaker implant.
* Inclusion in another trial which may influence the results of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Estimated)
Dates: Start 2024-07-12 (Actual); Primary Completion 2027-01-12 (Estimated); Study Completion 2027-01-12 (Estimated)

PRIMARY OUTCOMES:
Pacing-induced cardiomyopathy | 12 months
  Decrease in the left ventricular ejection fraction (LVEF) by >10% as compared to the LVEF before pacemaker implant and final LVEF<45%.

SECONDARY OUTCOMES:
LVEF during follow-up | 12 months
  To compare the mean or median (depending on distribution) LVEF before and one year after pacemaker implant in the two groups.
Mitral and tricuspid regurgitation | 12 months
  To compare the degree of mitral and tricuspid regurgitation before and one year after pacemaker implant in the two groups.
New York Heart Association (NYHA) class | 12 months
  To compare the NYHA class one year after pacemaker implant in the two groups.
Brain Natriuretic Peptide levels | 12 months
  To compare the N-terminal pro-B-type natriuretic peptide (NT-proBNP) levels one year after pacemaker implant in the two groups.
heart failure | 12 months
  Comparison of heart failure (HF) events in the first year after pacemaker implant in the two groups. HF events will be: hospitalizations for heart failure, emergency department or day-hospital visits for heart failure, heart failure symptoms requiring the initiation of diuretic therapy.

OTHER OUTCOMES:
Complications | 12 months
  Complications related to the ventricular lead

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Di Marco, MD, PhD, Principal Investigator — IDIBELL and Hospital Universitario de Bellvitge
Locations (6):
- Spain (6):
  - Hospital Vall d'Hebrón, Barcelona
  - Hospital General Universitario de Castellón, Castellon
  - Hospital Virgen de las Nieves, Granada
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat
  - Hospital La Fe, Valencia
  - Hospital Lozano Blesa, Zaragoza

IPD SHARING:
Plan to Share IPD: Yes
The study protocol and the informed consent form will be available upon request during the whole duration of the study.
Supporting Information: Study Protocol, ICF
Time Frame: During the whole duration of the study
Access Criteria: Request to the principal investigator.